CLINICAL TRIAL: NCT01757704
Title: Factors Responsible for the Effectiveness of the Lund Technique for De-airing Following Open Left Heart Surgery.
Brief Title: Factors Responsible for the Effectiveness of the Lund De-airing Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Bansi Lal Koul, Med dr. Ph. D., Lund University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BKML-003
Record Dates: First submitted 2012-09-22; First posted 2012-12-31 (Estimated); Results first posted 2013-12-06 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Complication of Surgical Procedure
Keywords: Cardiac de-airing; Air emboli; Trans-cranial Echo-Doppler; Intraoperative Trans-esophageal Echocardiography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open pleurae & conventional filling of heart (Experimental): In this group both pleurae will be opened and the ventilator disconnected during cardiopulmonary bypass to ensure bilateral pulmonary collapse. However, after completion of the left heart procedure, the heart will be filled with blood actively from the heart-lung machine and manual de-airing performed in a conventional manner and de-airing monitored by intraoperative trans-esophageal echocardiography (TEE). After de-airing is complete and patient has been weaned off the cardiopulmonary bypass the residual air in the left heart will be quantitatively assessed by TEE and Trans-cranial Echo-Doppler (TCD) over a period of 10 minutes.
  Interventions: Procedure: Open pleurae & conventional filling of heart
- Intact pleurae & staged filling of heart (Experimental): In this group both pleurae will be left intact and the ventilator disconnected during cardiopulmonary bypass. After completion of the left heart procedure, the heart will be filled with blood actively from the heart-lung machine in a staged manner after adequate cardiac contraction has been established. De-airing will be obtained by active cardiac contraction and staged mechanical ventilation and de-airing monitored by intraoperative trans-esophageal echocardiography (TEE). After de-airing is deemed complete and patient has been weaned off the cardiopulmonary bypass (CPB) the residual air in the left heart will be quantitatively assessed by TEE and Trans-cranial Echo-Doppler (TCD) over a period of 10 minutes.
  Interventions: Procedure: Intact pleurae & staged filling of heart

INTERVENTIONS:
Procedure: Open pleurae & conventional filling of heart — After completion of the left heart surgery, the heart will be actively filled with blood from the cardiopulmonary bypass circuit and lungs fully ventilated with positive end-expiratory pressure to flush out all air trapped in the lung veins and left heart. When there is no more visible air seen on Trans-esophageal echocardiography, the patient is weaned from cardiopulmonary bypass.
  Other Names: Cardiac de-airing; Cardiac venting
  Arms: Open pleurae & conventional filling of heart
Procedure: Intact pleurae & staged filling of heart — After the end of the left heart surgery, the heart is gradually filled with blood from the cardiopulmonary bypass circuit. Cardiac contractions fill the lungs with blood til no more air is seen in left heart on Trans-esophageal Echocardiography. Thereafter the lungs are ventilated with 50% of the estimated lung minute volume and 5 cm positive end-expiratory pressure and cardiac filling and de-airing continued. If no air is seen in the left heart full ventilation is started and the patient is weaned from cardiopulmonary bypass.
  Other Names: Cardiac de-airing; Cardiac venting
  Arms: Intact pleurae & staged filling of heart

SUMMARY:
The Lund de-airing technique is employed for cardiac de-airing in open left heart surgery. It consists of two main elements namely, opening of both pleura after the patient is on CPB (cardiopulmonary bypass)and disconnection of the ventilator before opening the left heart to ensure bilateral pulmonary collapse and a staged filling of the heart at termination of the CPB. The aim of this study is to analyze in a randomized manner two groups of patients to establish if one or both components are of primary importance for the effectiveness of the de-airing technique.

DETAILED DESCRIPTION:
Patients planned for open left heart surgery, mainly aortic valve replacement, will be included in the study. Patients with aortic valve replacement and concomitant coronary artery bypass with vein grafts only can also be included.

Exclusion criteria are; significant chronic obstructive pulmonary disease/emphysema, significant (>50%)carotid artery disease, need of concomitant internal mammary harvesting, prior cardiac or pulmonary surgery, pulmonary adhesions preventing pulmonary collapse, previous radiation to the chest and prior severe chest trauma. Intraoperative exclusion criteria are; failure to obtain adequate bilateral Trans-cranial Echo-Doppler signals from the medial cerebral arteries, finding of adherent pleurae and accidental opening of the pleurae.

Twenty patients will be randomized to two groups:

Group I: Intact pleura bilaterally, disconnection of the ventilator during cardiopulmonary bypass (CPB), followed by staged filling of the heart.

Group II: Open pleura bilaterally, disconnection of the ventilator during cardiopulmonary bypass to ensure bilateral pulmonary collapse followed by conventional filling of the heart.

Data will be compared to a third historical control group, consisting of ten patients with open pleurae with the ventilator disconnected followed by staged filling of the heart.

Primary outcomes:

* Duration of the de-airing procedure from the release of the aortic cross clamp to finished de-airing.
* Air microemboli to the brain registered on-line as gaseous microembolic signals on Trans-cranial Echo-Doppler (TCD). The sum of signals from the right and left middle cerebral artery are registered during the following time periods; from the release of the aortic cross clamp to start of cardiac ejection, from cardiac ejection to finished de-airing, and during ten minutes after finished de-airing.
* Magnitude of residual air emboli in the heart after finished de-airing as monitored by Trans-esophageal Echocardiography (TEE) with a Three-chamber view. The severity of residual air is classified in four grades after the appearance of visible air on TEE in left atrium (LA), left ventricle (LV) and aortic root (AO)as follows; Grade 0: no residual air, grade I: gas emboli detected in one of three anatomic areas during one cardiac cycle, grade II: gas emboli detected simultaneously in two of three anatomic areas during one cardiac cycle; grade III: gas emboli detected in all three anatomic areas during one cardiac cycle.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for aortic valve replacement with or without coronary vein bypass grafts

Exclusion Criteria:

* Significant chronic obstructive pulmonary disease and emphysema
* Previous history of thoracic or cardiac surgery
* Patients requiring internal mammary artery harvesting
* Unilateral or bilateral pulmonary adhesions to chest wall
* Previous radiation to the chest

Intraoperative Exclusion Criteria:

* Inability to obtain adequate bilateral Trans-cranial Echo-doppler signals
* Adherent pleurae
* Accidental opening of the pleurae

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bansi Koul, MD, PhD, Principal Investigator — Cardiothoracic Surgery, Skåne University Hospital Lund, Sweden
Locations (1):
- Lund University, Lund, Skåne County, Sweden

REFERENCES:
- [Background] Al-Rashidi F, Blomquist S, Hoglund P, Meurling C, Roijer A, Koul B. A new de-airing technique that reduces systemic microemboli during open surgery: a prospective controlled study. J Thorac Cardiovasc Surg. 2009 Jul;138(1):157-62. doi: 10.1016/j.jtcvs.2009.02.037. PMID 19577073
- [Background] Al-Rashidi F, Landenhed M, Blomquist S, Hoglund P, Karlsson PA, Pierre L, Koul B. Comparison of the effectiveness and safety of a new de-airing technique with a standardized carbon dioxide insufflation technique in open left heart surgery: a randomized clinical trial. J Thorac Cardiovasc Surg. 2011 May;141(5):1128-33. doi: 10.1016/j.jtcvs.2010.07.013. Epub 2010 Sep 3. PMID 20817209

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who were scheduled at the Department of Cardiothoracic Surgery, anesteshia and intensive care at Skane University Hospital for elective open left sided heart surgery were eligible for inclusion. Recruitment started in september 2012 and ended in june 2013.
Pre-assignment Details: In this study a total of 4 participants did not complete due to intraoperative exclusion criteria only possible to detect after start of the surgical procedure (adherant lung, accidental pleural opening, TCD signal insufficient). Enrollment and randomization continued until 10 patients in each arm were included and satisfied protocol criteria.
Groups:
- Intact Pleurae & Staged Filling of Heart: In this group both pleurae will be left intact and the ventilator disconnected during cardiopulmonary bypass. After completion of the left heart surgery, the heart will be filled with blood actively from the heart-lung machine in a staged manner after adequate cardiac contraction has been established. De-airing will be obtained by active cardiac contraction and staged mechanical ventilation and de-airing monitored by intraoperative trans-esophageal echocardiography (TEE). After de-airing is deemed complete and patient has been weaned off the cardiopulmonary bypass (CPB) the residual air in the left heart will be quantitatively assessed by TEE and Trans-cranial Echo-Doppler (TCD) over a period of 10 minutes.
  Intact pleurae & staged filling of heart : After the end of the left heart surgery, the heart is gradually filled with blood from the cardiopulmonary bypass circuit. Cardiac contractions fill the lungs with blood til no more air is seen in left heart on Trans-esophageal Echocar
- Open Pleurae & Conventional Filling of Heart: In this group both pleurae will be opened and the ventilator disconnected during cardiopulmonary bypass to ensure bilateral lung collapse. However, after completion of the left heart procedure, the heart will be filled with blood actively from the heart-lung machine and manual de-airing performed in a conventional manner and de-airing monitored by intraoperative trans-esophageal echocardiography (TEE). After de-airing is complete and patient has been weaned off the cardiopulmonary bypass the residual air in the left heart will be quantitatively assessed by TEE and Trans-cranial Echo-Doppler (TCD) over a period of 10 minutes.
  Open pleurae & conventional filling of heart : After completion of the left heart surgery, the heart will be actively filled with blood from the cardiopulmonary bypass circuit and lungs fully ventilated with positive end-expiratory pressure to flush out all air trapped in the lung veins and left heart. When there is no more visible air seen on trans-esophag
Period: Overall Study
Arm/Group | Intact Pleurae & Staged Filling of Heart | Open Pleurae & Conventional Filling of Heart
Started | 11 (One patient was excluded at start of surgery due to opening of the pleurae during sternotomy.) | 13 (Two patients excluded intraoperatively due to failure to obtain TCD signals and one due to adhesion.)
Completed | 10 | 10
Not Completed | 1 | 3
Not completed — Protocol Violation | 1 | 3

BASELINE CHARACTERISTICS:
Population: Only participants that did not fulfill intraoperative exclusion criteria continued throughout the study according to the study protocol and were included in baseline data analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intact Pleurae & Staged Filling of Heart | Open Pleurae & Conventional Filling of Heart | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (12.5) | 71.1 (11.5) | 70.2 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  Sweden | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Assessment of Air Embolism to the Brain After Completion of Open Left Heart Surgery
Description: Cerebral air emboli will be assessed quantitatively by On-line counting of gaseous microembolic signals (MES) by Trans-cranial Echo-Doppler (TCD) monitoring of the right and left middle cerebral artery. The sum of the gaseous microembolic signals registered from the right and left middle cerebral artery will be reported.
Time Frame: Time from the release of the aortic crossclamp to cardiac ejection, an average of 10-15 minutes
Measure: Median (Inter-Quartile Range); unit: Air microemboli
Arm/Group | Intact Pleurae & Staged Filling of Heart | Open Pleurae & Conventional Filling of Heart
Number analyzed (Participants) | 10 | 10
Air microemboli | 49 [44 to 113] | 46 [43 to 69]

2. Primary Outcome: Quantitative Assessment of Air Embolism to the Brain After Completion of Open Left Heart Surgery
Description: as for outcome 1
Time Frame: Time from cardiac ejection to finished de-airing, an average of 5-10 minutes
Measure: Median (Inter-Quartile Range); unit: Air microemboli
Arm/Group | Intact Pleurae & Staged Filling of Heart | Open Pleurae & Conventional Filling of Heart
Number analyzed (Participants) | 10 | 10
Air microemboli | 71 [32 to 281] | 28 [14 to 41]

3. Primary Outcome: Quantitative Assessment of Air Embolism to the Brain After Completion of Open Left Heart Surgery
Description: as for outcome 1
Time Frame: Period of ten minutes after finished de-airing
Measure: Median (Inter-Quartile Range); unit: Air microemboli
Arm/Group | Intact Pleurae & Staged Filling of Heart | Open Pleurae & Conventional Filling of Heart
Number analyzed (Participants) | 10 | 10
Air microemboli | 65 [38 to 210] | 9 [6 to 36]
Statistical Analysis 1: Comparison: Intact Pleurae & Staged Filling of Heart vs Open Pleurae & Conventional Filling of Heart; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney); Median Difference (Net) = 56

4. Primary Outcome: Participants With <=Grade I Air Emboli as Assessed by Trans-esophageal Echocardiography (TEE) After Finished De-airing.
Description: The severity of residual air emboli in three anatomic areas; left atrium, left ventricle and aortic root, is assessed by Trans-esophageal Echocardiography (TEE) and classified in grade 0-3 as follows, Grade o: no residual air; grade I: gas emboli detected in one of three anatomic areas during one cardiac cycle; grade II: gas emboli detected simultaneously in two of three anatomic areas during one cardiac cycle; grade III: gas emboli detected simultaneously in all three anatomic areas during one cardiac cycle.
Time Frame: 0-3 minutes after finished de-airing
Measure: Number; unit: Participants
Arm/Group | Intact Pleurae & Staged Filling of Heart | Open Pleurae & Conventional Filling of Heart
Number analyzed (Participants) | 10 | 10
Participants | 3 | 10

5. Primary Outcome: Participants With <=Grade I Air Emboli as Assessed by Trans-esophageal Echocardiography (TEE) After Finished De-airing.
Description: as for outcome 4
Time Frame: 3-6 minutes after finished de-airing
Measure: Number; unit: Participants
Arm/Group | Intact Pleurae & Staged Filling of Heart | Open Pleurae & Conventional Filling of Heart
Number analyzed (Participants) | 10 | 10
Participants | 6 | 10

6. Primary Outcome: Participants With <=Grade I Air Emboli as Assessed by Trans-esophageal Echocardiography (TEE) After Finished De-airing.
Description: as for outcome 4
Time Frame: 6-10 minutes after finished de-airing
Measure: Number; unit: Participants
Arm/Group | Intact Pleurae & Staged Filling of Heart | Open Pleurae & Conventional Filling of Heart
Number analyzed (Participants) | 10 | 10
Participants | 9 | 10

7. Primary Outcome: Duration of the De-airing Procedure
Description: The de-airing procedure is deemed completed when the Trans-esophageal Echocardiography (TEE) no longer visualizes air emboli in the heart Chambers. The duration is likely to vary between individuals and reflects the complexity of the de-airing procedure.
Time Frame: Time from release of aortic crossclamp to finished de-airing
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Intact Pleurae & Staged Filling of Heart | Open Pleurae & Conventional Filling of Heart
Number analyzed (Participants) | 10 | 10
Minutes | 14 [10 to 20] | 8.5 [6 to 12]

ADVERSE EVENTS:
Time Frame: Postoperative hospital stay, an average of 7 Days.
Description: Participants medical charts were studied to find reported signs of postoperative neurological dysfunction that included clinical signs of stroke or transient neurological deficit. Transient neurological dysfunction was defined as severe confusion, agitation or hallucinations.
Arm/Group | Intact Pleurae & Staged Filling of Heart | Open Pleurae & Conventional Filling of Heart
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intact Pleurae & Staged Filling of Heart (N=10) | Open Pleurae & Conventional Filling of Heart (N=10)
cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intact Pleurae & Staged Filling of Heart (N=10) | Open Pleurae & Conventional Filling of Heart (N=10)
cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) — Confirmed by cerebral CT scan on postoperative day 2.

LIMITATIONS AND CAVEATS:
This study is a small single center study. Though randomized and controlled, the surgeon and anesthesiologist were not blinded to which arm a participant belonged to during the course of surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes